CLINICAL TRIAL: NCT04601467
Title: PASSIvation of Vulnerable Plaque With AZD5718 in AcuTe Coronary syndromE
Acronym: PASSIVATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early on 14th September 2023 by the main funding company because of financial futility. We were able to enroll 243 of the initial planned 360 participants and randomised 209 participants of the intial planned 286.
Sponsor: National University Heart Centre, Singapore (Other)
Collaborators: AstraZeneca (Industry); University of Otago (Other)
Responsible Party: Principal Investigator, Mark Chan, Associate Professor, National University Heart Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/
Record Dates: First submitted 2020-09-11; First posted 2020-10-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Myocardial Infarction; Computed Tomography Coronary Angiography
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — AZD5718

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: CT coronary angiogram core laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD5718 (Experimental): Patients will receive once daily oral dose of AZD5718 for 12 months
  Interventions: Drug: AZD5718
- Placebo (Placebo Comparator): Patients will receive once daily oral dose of placebo matched to AZD5718 for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5718 — Oral dose of AZD5718 (tablet) once daily for 12 months
  Arms: AZD5718
Drug: Placebo — Oral dose of matching placebo (tablet) once daily for 12 months
  Arms: Placebo

SUMMARY:
This is a multi-center study conducted at 8 sites in 2 countries (Singapore, New Zealand). Patients with an acute myocardial infarction (AMI) were randomized in a ratio of 1:1 ratio to receive AZD5718 (Atuliflapon) 125 mg or placebo for 12 months to assess the efficacy of AZD5718 to prevent coronary plaque progression as measured on serial computer tomographic coronary angiography.

DETAILED DESCRIPTION:
PASSIVATE is a randomized, double-blind, placebo-controlled Phase IIa trial that investigates how 12 months of treatment with AZD5718 modifies coronary plaque volume. Patients with recent STEMI or NSTEMI will receive an additional oral dose of AZD5718 (or placebo) once daily to standard clinical care for 12 months. The primary hypothesis being tested in PASSIVATE is that 12 months of treatment with AZD5718 attenuates the progression of non-calcified plaque (NCP) volume on serial computed tomography coronary angiography (CTCA) studies.

Patients who gave consent (within 60 days after their index event) will undergo a CTCA scan and start treatment (AZD5718 or Placebo). The treatment duration will be 12 months. During the treatment period, patients will come to the clinic for follow-ups. At 12 months (end treatment), the patients will undergo their 2nd CTCA scan. A follow-up visit will be performed 4 weeks after the last dose in order to ensure the safety and well-being of the patients.

ELIGIBILITY:
Inclusion Criteria:

* hospitalised for STEMI or non-STEMI, as defined by the 4th universal definition of MI
* underwent coronary angiography during the index hospitalisation showing at least one epicardial coronary artery with ≥50% stenosis and a 2nd epicardial coronary artery with ≥20% stenosis on the coronary angiogram
* Body Mass Index (BMI) ≥18 to ≤40 kg/m2
* White Blood Cell count ≥ 7.0 X 103/uL during admission

Exclusion Criteria:

* Prior coronary artery bypass grafting (CABG)
* CABG planned within 12 months of admission
* Known history of drug or alcohol abuse within 5 years of screening
* History of QT prolongation associated with other medications that required discontinuation of that medication
* Congenital long QT syndrome
* Systolic blood pressure persistently <90 mm Hg or HR<40 beats per minute at time of enrolment
* ALT >2 x ULN, cirrhosis, recent hepatitis, or positive screening test for hepatitis B (hepatitis B surface antigen) or other viral hepatitis
* Uncontrolled Type 1 or Type 2 DM defined as HbA1c >10% or 74.9 mmol/mol (by IFCC)
* Any planned coronary revascularisation, valve surgery, or cardiac resynchronisation within 7 months after randomisation
* Any concomitant medications known to be associated with Torsades de Pointes or potent inducers of cytochrome P450 3A4 (CYP3A4)
* Planned treatment with zileuton, leukotriene receptor antagonists (e.g., montelukast) during trial
* Participated in another interventional clinical study with an investigational pharmaceutical product during the last 3 months
* Known hypersensitivity to drugs with a similar chemical structure or class of study drugs or any of the excipients of the product
* Known conditions that either increase the risk of performing the CT or make the procedure technically impractical
* No severe asthma attack that require emergency treatment or hospitalisation in the past 6 months
* Had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated), and/or had a confirmed case of COVID-19 within 4 weeks of Screening Visit

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Change in noncalcified coronary artery plaque volume (NCPV) | Baseline (before treatment) and after 12 months of treatment
  Percent change in NCPV (in mm3), as assessed by CT coronary angiography, from baseline (before treatment) to after 12-month of treatment

SECONDARY OUTCOMES:
Change in CT peri vascular (coronary) adipose tissue (PVAT) | Baseline (before treatment) and after 12 months of treatment
  To assess whether AZD5718 reduces coronary inflammation
Change in total plaque volume (mm3) | Baseline (before treatment) and after 12 months of treatment
  Percent change in total plaque volume (in mm3), as assessed by CT coronary angiography, from baseline (before treatment) to after 12-month of treatment
Echocardiographic assessment: Change in left ventricular ejection fraction (LVEF) | Baseline (before treatment) and after 12 months of treatment
  Percent change in LVEF (%), as assessed by 2D echocardiography, from baseline (before treatment) to after 12-month of treatment
Change in levels of urinary LTE4 (u-LTE4) | 12 months
  To assess the pharmacodynamics (PD) effect of AZD5718 by assessment of u-LTE4 in AMI patients

OTHER OUTCOMES:
Change in low attenuation plaque burden | Baseline (before treatment) and after 12 months of treatment
  Percent change in low attenuation (<30 HU) plaque volume (mm3), as assessed by CT coronary angiography, from baseline (before treatment) to after 12-month of treatment
Change in plasma hs-CRP concentration | Baseline (before treatment) and after 12 months of treatment
  To assess the changes in circulating hs-CRP concentrations from baseline (before treatment) to after 12-month of treatment
Echocardiographic assessment: Change in LV global longitudinal strain | Baseline (before treatment) and after 12 months of treatment
  Percent change in LV global longitudinal strain, as assessed by 2D echocardiography, from baseline (before treatment) to after 12-month of treatment
Echocardiographic assessment: Change in global circumferential strain | Baseline (before treatment) and after 12 months of treatment
  Percent change in global circumferential strain, as assessed by 2D echocardiography, from baseline (before treatment) to after 12-month of treatment
Echocardiographic assessment: Change in longitudinal early diastolic strain rate | Baseline (before treatment) and after 12 months of treatment
  Percent change in longitudinal early diastolic strain rate, as assessed by 2D echocardiography, from baseline (before treatment) to after 12-month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chan, Principal Investigator — National University Heart Centre, Singapore; Derek Hausenloy, Principal Investigator — National Heart Centre Singapore; A. Mark Richards, Study Chair — National University Heart Centre, Singapore
Locations (8):
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Christchurch Heart Institute (CHI), Christchurch
- Singapore (6):
  - Changi General Hospital (CGH), Singapore
  - Khoo Teck Puat Hospital (KTPH), Singapore
  - National Heart Centre Singapore (NHCS), Singapore
  - National University Heart Centre, Singapore (NUHCS), Singapore
  - Ng Teng Fong General Hospital (NTFGH), Singapore
  - Tan Tock Seng Hospital (TTSH), Singapore

IPD SHARING:
Plan to Share IPD: Yes
We will share anonmyised IPD upon reasonable request from academic investigators employed by universities and/or healthcare organisations to the study PIs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date and end date will be specified upon publication of the primary trial results
Access Criteria: Only investigators employed by universities or healthcare organisations upon reasonable request to the study PIs.
URL: https://medicine.nus.edu.sg/trp/cardiovascular-disease/flagship-projects/passivate/

REFERENCES:
- [Background] Ericsson H, Nelander K, Lagerstrom-Fermer M, Balendran C, Bhat M, Chialda L, Gan LM, Heijer M, Kjaer M, Lambert J, Lindstedt EL, Forsberg GB, Whatling C, Skrtic S. Initial Clinical Experience with AZD5718, a Novel Once Daily Oral 5-Lipoxygenase Activating Protein Inhibitor. Clin Transl Sci. 2018 May;11(3):330-338. doi: 10.1111/cts.12546. Epub 2018 Mar 8. PMID 29517132
- [Background] Pettersen D, Broddefalk J, Emtenas H, Hayes MA, Lemurell M, Swanson M, Ulander J, Whatling C, Amilon C, Ericsson H, Westin Eriksson A, Granberg K, Plowright AT, Shamovsky I, Dellsen A, Sundqvist M, Nagard M, Lindstedt EL. Discovery and Early Clinical Development of an Inhibitor of 5-Lipoxygenase Activating Protein (AZD5718) for Treatment of Coronary Artery Disease. J Med Chem. 2019 May 9;62(9):4312-4324. doi: 10.1021/acs.jmedchem.8b02004. Epub 2019 Mar 26. PMID 30869888